CLINICAL TRIAL: NCT02892253
Title: Parathyroid Autofluorescence Visualization in Thyroid Surgery: Impact on Postoperative Hypocalcemia. A Randomized Controlled Trial
Brief Title: Parathyroid Autofluorescence Visualization in Thyroid Surgery: Impact on Postoperative Hypocalcemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Fares BENMILOUD, MD, Hôpital Européen Marseille
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-A-000549-42ParaFluo2
Record Dates: First submitted 2016-09-01; First posted 2016-09-08 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Hypocalcemia
Keywords: postoperative hypocalcemia; near infrared imaging; parathyroid autofluorescence
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIR+ group (Experimental): Patients who undergo conventional total thyroidectomy (TT)+/- lymph node dissection (LND).
  Parathyroid identification was done with the use of NIR (intervention group, NIR+ group)
  Interventions: Device: Near Infrared Camera (NIR)
- NIR- group (No Intervention): Patients who undergo conventional total thyroidectomy (TT)+/- lymph node dissection (LND) without the use of NIR - parathyroid identification was done by naked eye only (no intervention group, NIR- group)

INTERVENTIONS:
Device: Near Infrared Camera (NIR) — Surgical field is examined with NIR, during a few minutes (<5') with room lights switched off, to avoid parasite lights, then open thyroidectomy is resumed conventionally. Real-time images, evocative of autofluorescent parathyroids, are checked visually. NIR consists of a 750 nm class 1 laser excitation, with a power <20mW/cm2 (5 times less than the limit of 100mw/cm2, fixed by the international standard IEC 60601-2-41). It is provided by the Fluobeam® camera, which is inserted into a sterile cover and hold at a 15-20 cm distance from the patient. The system has an FDA 510(k) authorization for clinical use in parathyroid surgery and a European Community certification (Class 2A device).
  Other Names: Fluobeam® system (Fluoptics®, Grenoble, France)
  Arms: NIR+ group

SUMMARY:
This Multicenter, Randomized Controlled Trial evaluates the clinical impact of parathyroid autofluorescence visualization using near infrared light (NIR) during total thyroidectomy (TT). It compares patients who undergo TT associated or not with lymph node dissection (LND) with NIR vs without NIR use during surgery.

DETAILED DESCRIPTION:
Total thyroidectomy (TT) is responsible for postoperative hypocalcemia in 20-30% of patients, which is definitive in 1-4% of operated patients (1). This complication is mainly due to surgery-induced parathyroid dysfunction, which could be improved by a better intraoperative identification of the parathyroids. Intraoperative parathyroid auto-fluorescence visualization (without any dye injection) using near infrared light (NIR) is an emerging technique, which allows correct identification of normal parathyroids in almost all cases (2), but the clinical impact of NIR is unknown.

The aim of this prospective, comparative randomized study, is to compare 2 groups of patients: patients operated with NIR (NIR+) vs patients operated without NIR (NIR-).

The main objective of this study is to assess the impact of intraoperative use of NIR camera on postoperative hypocalcemia. Secondary objectives are to assess the impact of NIR on the visualization, autotransplantation and inadvertent resection rates during TT.

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for one-stage total thyroidectomy, associated or not to lymph node dissection (TT +/- LND).

Exclusion Criteria:

* Combined parathyroid and thyroid disease (including patients with enlarged parathyroids incidentally found during surgery and resected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Postoperative hypocalcemia | 6 months
  Postoperative day 1 and day 2 corrected calcemia (hypocalcemia when calcemia <2mmol/l). If hypocalcemia, calcium is measured at 1 month and 6 months

SECONDARY OUTCOMES:
Number of identified parathyroids | immediate (intraoperative)
  identified by naked eye
Number of autotransplanted parathyroids | immediate (intraoperative)
  when parathyroids cannot be left in situ, they are fragmented and reinserted in a sterno-cleido-mastoid muscle
Number of inadvertently resected parathyroids | delayed (10 days)
  when parathyroid tissue is found on thyroid specimen (reported on pathology report)

CONTACTS AND LOCATIONS:
Overall Officials: BENMILOUD Fares, MD, Principal Investigator — Hopital Europeen de Marseille; BIDAUT Wahiba, Senior CRA, Study Chair — Hopital Europeen de Marseille; REBAUDET Stanislas, MD, Study Chair — Hopital Europeen de Marseille; PENARANDA Guillaume, Study Chair — Laboratoire Alphabio
Locations (3):
- France (3):
  - Hopital Europeen, Marseille
  - Hôpital Saint Joseph Marseille, Marseille
  - Hopital La Pitie Salpetriere, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duclos A, Peix JL, Colin C, Kraimps JL, Menegaux F, Pattou F, Sebag F, Touzet S, Bourdy S, Voirin N, Lifante JC; CATHY Study Group. Influence of experience on performance of individual surgeons in thyroid surgery: prospective cross sectional multicentre study. BMJ. 2012 Jan 10;344:d8041. doi: 10.1136/bmj.d8041. PMID 22236412
- [Background] McWade MA, Sanders ME, Broome JT, Solorzano CC, Mahadevan-Jansen A. Establishing the clinical utility of autofluorescence spectroscopy for parathyroid detection. Surgery. 2016 Jan;159(1):193-202. doi: 10.1016/j.surg.2015.06.047. Epub 2015 Oct 9. PMID 26454675
- [Derived] Benmiloud F, Godiris-Petit G, Gras R, Gillot JC, Turrin N, Penaranda G, Noullet S, Chereau N, Gaudart J, Chiche L, Rebaudet S. Association of Autofluorescence-Based Detection of the Parathyroid Glands During Total Thyroidectomy With Postoperative Hypocalcemia Risk: Results of the PARAFLUO Multicenter Randomized Clinical Trial. JAMA Surg. 2020 Feb 1;155(2):106-112. doi: 10.1001/jamasurg.2019.4613. PMID 31693081